CLINICAL TRIAL: NCT05483049
Title: Prevalence of Significant Liver Fibrosis and Inflammation in Chronic HBV Infected Patients in Grey Zone
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, WANG HUI, PROFESSOR, Ruijin Hospital
Other Study IDs: liver injury-grey zone
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — liver biopsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- grey zone 1: HBeAg (+), HBV DNA >20 but < 10000000IU/mL, ALT ≤40 U/L
- grey zone 2: HBeAg (-), HBV DNA > 2000 IU/mL, ALT ≤40 U/L

SUMMARY:
To explore whether normal alanine aminotransferase (ALT) is associated with liver injury in a cohort of hepatitis B virus (HBV) infected patients in grey zone

DETAILED DESCRIPTION:
Hepatitis B is caused by HBV infection, which can progress to chronic HBV infection after 6 months. HBV infection is a global public health problem, which can affect liver function and even threaten life health. HBV infection is worldwide prevalent, but the infection rate varies greatly in different regions. According to World Health Organization (WHO), there are about 257 million chronic HBV infections worldwide. The western Pacific region and Africa are the most prevalent regions of HBV, with the adult infection rate of 6.2% and 6.1% respectively. Most of Asia is a medium-high epidemic area 1. In 2014, Center for Disease Control and Prevention (CDC) conducted a serological epidemiological survey on hepatitis B among the population aged 1-29 in China, and the results showed that the prevalence rate of HBsAg in the population aged 1-4, 5-14 and 15-29 was 0.32%, 0.94% and 4.38%, respectively. It is estimated that the prevalence of HBsAg in the general population of China is 5-6%, and there are about 70 million chronic HBV infections, among which there are about 20-30 million chronic hepatitis B (CHB) patients. Chronic HBV infection increases the risk of liver fibrosis and hepatocellular carcinoma (HCC). The annual incidence of cirrhosis is 2-10% in CHB patients without antiviral therapy, and the annual incidence of HCC in patients with cirrhosis is 3-6%2.

The China 2019 Prevention and Treatment Guidelines of Chronic Hepatitis B recommend that patients with positive HBV DNA and elevated ALT, and those above 30 years old with family history of liver cirrhosis or HCC should initiate antiviral treatment, after ruling out other potential causes. However, the guideline did not identify the specific reference value of upper limit of normal for ALT, neither with cut off value of HBV detection. In addition, there is no clear definition of 'family history'. So, the fuzzy boundaries in the HBV guidelines may cause confusion when providing treatment recommendations in clinical practice and the value of this study would contribute to solve this kind of problems.

In a recently published study this year, 432 CHB patients who had liver biopsy in Ruijin Hospital during 2011-2017 were reviewed. So based on this, In the present study, we estimated a sample size of 600.Chronic HBV infected patients from 4 sites who underwent liver biopsy between 2008 and 2020.12 will be enrolled.

Previous studies have shown that a high proportion of HBV-infected patients with normal ALT have significant liver injury, including significant inflammation or fibrosis, and even cirrhosis.

And studies also show that treatment naive patients with normal ALT, either HBeAg-positive or HBeAg-negative, have a higher risk of developing HCC and even death than those in immune-active patients who received antiviral treatment (AVT). Therefore, early identification of patients with normal ALT but with significant liver inflammation or fibrosis is crucial.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve
* serum HBsAg positive for >6 months
* Grey zone 1: HBeAg (+), HBV DNA >20 but < 107IU/mL, ALT ≤40 U/L
* Grey zone 2: HBeAg (-), HBV DNA > 2000 IU/mL, ALT ≤40 U/L

Exclusion Criteria:

* Co-infection with HCV, HDV or HIV
* decompensated cirrhosis
* other chronic liver diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An estimated 600 chronic HBV infected patients who underwent liver biopsy between Jan, 2008 and December, 2021 will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of significant liver fibrosis. | from Jan, 2008 to December, 2021
  Prevalence of significant liver fibrosis (G≥2) in patients in all patients.
Prevalence of significant liver inflammation. | from Jan, 2008 to December, 2021
  Prevalence of significant liver inflammation (S≥2) in patients in all patients.

SECONDARY OUTCOMES:
Prevalence of significant liver fibrosis in different age group in grey zone 1. | from Jan, 2008 to December, 2021
  Prevalence of significant liver fibrosis (G≥2) in different age group (10 years old per group) in patients in grey zones 1.
Prevalence of significant liver inflammation in different age group in grey zone 1. | from Jan, 2008 to December, 2021
  Prevalence of significant liver inflammation (S≥2) in different age group (10 years old per group) in patients in grey zones 1.
Prevalence of significant liver fibrosis in different age group in grey zone 2. | from Jan, 2008 to December, 2021
  Prevalence of significant liver fibrosis (G≥2) in different age group (10 years old per group) in patients in grey zones 2.
Prevalence of significant liver inflammation in different age group in grey zone 2. | from Jan, 2008 to December, 2021
  Prevalence of significant liver inflammation (S≥2) in different age group (10 years old per group) in patients in grey zones 2.
Prevalence of significant liver fibrosis at different ALT level in grey zone 1. | from Jan, 2008 to December, 2021
  Prevalence of significant liver fibrosis (G≥2)at different ALT level (low normal level 0-25 U/L for women and 0-35 U/L for men, high normal level 26-40 U/L for women and 36-40 U/L for men) in patients in grey zones 1.
Prevalence of significant liver inflammation at different ALT level in grey zone 1. | from Jan, 2008 to December, 2021
  Prevalence of significant liver inflammation (S≥2) at different ALT level (low normal level 0-25 U/L for women and 0-35 U/L for men, high normal level 26-40 U/L for women and 36-40 U/L for men) in patients in grey zones 1.
Prevalence of significant liver fibrosis at different ALT level in grey zone 2. | from Jan, 2008 to December, 2021
  Prevalence of significant liver fibrosis (G≥2)at different ALT level (low normal level 0-25 U/L for women and 0-35 U/L for men, high normal level 26-40 U/L for women and 36-40 U/L for men) in patients in grey zones 2.
Prevalence of significant liver inflammation at different ALT level in grey zone 2. | from Jan, 2008 to December, 2021
  Prevalence of significant liver inflammation (S≥2) at different ALT level (low normal level 0-25 U/L for women and 0-35 U/L for men, high normal level 26-40 U/L for women and 36-40 U/L for men) in patients in grey zones 2.
Prevalence of significant liver fibrosis at different DNA level in grey zone 1. | from Jan, 2008 to December, 2021
  Prevalence of significant liver fibrosis (G≥2) at different DNA level (log10 IU/mL per group) in patients in grey zones 1.
Prevalence of significant liver inflammation at different DNA level in grey zone 1. | from Jan, 2008 to December, 2021
  Prevalence of significant liver inflammation (S≥2) at different DNA level (log10 IU/mL per group) in patients in grey zones 1.
Prevalence of significant liver fibrosis at different DNA level in grey zone 2. | from Jan, 2008 to December, 2021
  Prevalence of significant liver fibrosis (G≥2) at different DNA level (log10 IU/mL per group) in patients in grey zones 2.
Prevalence of significant liver inflammation at different DNA level in grey zone 2. | from Jan, 2008 to December, 2021
  Prevalence of significant liver inflammation (S≥2) at different DNA level (log10 IU/mL per group) in patients in grey zones 2.
Prevalence of significant liver fibrosis with different family history of HCC in grey zone 1. | from Jan, 2008 to December, 2021
  Prevalence of significant liver fibrosis (G≥2) with different family history of HCC or liver cirrhosis (first degree relative, second and third degree relatives) in patients in grey zones 1.
Prevalence of significant liver inflammation with different family history of HCC in grey zone 1. | from Jan, 2008 to December, 2021
  Prevalence of significant liver inflammation (S≥2) with different family history of HCC or liver cirrhosis (first degree relative, second and third degree relatives) in patients in grey zones 1.
Prevalence of significant liver fibrosis with different family history of HCC in grey zone 2. | from Jan, 2008 to December, 2021
  Prevalence of significant liver fibrosis (G≥2) with different family history of HCC or liver cirrhosis (first degree relative, second and third degree relatives) in patients in grey zones 2.
Prevalence of significant liver inflammation with different family history of liver cirrhosis in grey zone 2. | from Jan, 2008 to December, 2021
  Prevalence of significant liver inflammation (S≥2) with different family history of HCC or liver cirrhosis (first degree relative, second and third degree relatives) in patients in grey zones 2.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wang, Principal Investigator — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: No